CLINICAL TRIAL: NCT06393062
Title: Gram Stain of the First Urine After Intraoperative Renal Puncture in Predicting the Systemic Inflammatory Response After Percutaneous Nephrolithotomy: A Prospective, Randomized Controlled Study
Brief Title: Gram Stain of the First Urine After Puncture in Percutaneous Nephrolithotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Bedreddin Kalyenci, Assistant professor doctor, Adiyaman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022/7-17
Record Dates: First submitted 2024-04-24; First posted 2024-05-01 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Percutaneous Nephrolithotomy
Keywords: fever; gram stain; percutaneous nephrolithotomy; Systemic inflammatory response syndrome (SIRS)
MeSH Terms: conditions — Fever; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Intervention Model Description: The patients included in the study were randomized by a block randomization method by an independent researcher, hidden from the patients and the responsible clinicians, using a computerized number tool.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gram staining (Experimental): Gram staining of post-puncture urine in percutaneous nephrolithotomy
  Interventions: Diagnostic Test: Gram staining of the first urine after intraoperative renal puncture to predict the systemic inflammatory response after percutaneous nephrolithotomy.
- control (No Intervention): non-intervention percutaneous nephrolithotomy

INTERVENTIONS:
Diagnostic Test: Gram staining of the first urine after intraoperative renal puncture to predict the systemic inflammatory response after percutaneous nephrolithotomy. — Gram staining of the first urine after intraoperative renal puncture to predict the systemic inflammatory response after percutaneous nephrolithotomy.
  Arms: Gram staining

SUMMARY:
In this study, investigators compared the systemic inflammatory responses after percutaneous nephrolithotomy (PCNL) patients who were given an expanded empirical antibiotic regimen based on the prediction of the possibility of bacteria identified by Gram staining the first urine after renal puncture and patients whose antibiotic regimen was not performed and whose antibiotic regimen was adjusted according to patient symptoms and culture results. Investigators aimed to test its diagnostic value in predicting and preventing complications.

ELIGIBILITY:
Inclusion Criteria:

* patients with an indication for percutaneous nephrolithotomy due to kidney stone disease.

Exclusion Criteria:

* under 18 years old,
* having an active urinary tract infection before surgery and positive urine cultures,
* Patients with bilateral kidney stones,
* DJ stent or nephrostomy placement,
* Solitary kidney stones,
* Bleeding disorders,
* impaired kidney function,
* a history of antibiotic use for any reason within 2 weeks before randomization were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Gram stain in predicting systemic inflammatory response after percutaneous nephrolithotomy. | immediately after the surgery
  Gram staining of urine after puncture to detect the presence of bacteria that are a possible source of infection according to the rate of gram-stained and non-gram-stained patients by microscopic examination.

SECONDARY OUTCOMES:
Change of antibiotic regimen after bacterial estimation of Gram stain | immediately after the surgery
  The percentage of patients whose antibiotic regimen was changed by estimating bacteria after Gram staining did not progress to systemic inflammatory response syndrome. Systemic inflammatory response criteria: temperature less than 36 °C or higher than 38 °C, heart rate more than 100 beats per minute, respiratory rate more than 20 per minute, leukocyte count greater than 12 × 10 up 9/L or 4 × 10 up 9/L less than L, systolic blood pressure falling below 90 mmHg, or diastolic blood pressure falling below 40 mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman University, Medicine of Faculty, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Patient clinical data before and after surgery
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: Data will be shared with all researchers conducting research on the prevention and detection of infectious consequences after percutaneous nephrolithotomy.